CLINICAL TRIAL: NCT02058264
Title: A Randomized, Double Blinded, Vehicle-Controlled Study to Evaluate the Safety and the Effect on Sweat Production of Topically Applied BBI-4000 in Subjects With Hyperhidrosis.
Brief Title: A Safety, Tolerability and Preliminary Efficacy Study of BBI-4000 in Subjects With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBI-4000-CL-101
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Low Strength BBI-4000 and Vehicle (Experimental)
  Interventions: Drug: BBI-4000
- High Strength BBI-4000 and Vehicle (Experimental)
  Interventions: Drug: BBI-4000

INTERVENTIONS:
Drug: BBI-4000

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and treatment effect of BBI-4000 when topically applied to subjects with axillary hyperhidrosis.

DETAILED DESCRIPTION:
This is a randomized, vehicle controlled, double blind study in subjects with axillary hyperhidrosis designed to assess the safety, tolerability and the effect on sweat production of topically applied BBI-4000 for 14 days.

Safety will be assessed though vital signs, physical exam, adverse events, local skin reactions and laboratory tests (blood chemistry and hematology).

Efficacy will be assessed though the gravimetrically measured sweat production and the Hyperhidrosis Disease Severity Score (HDSS).

Pharmacokinetic information will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female subjects from 18 to 45 years of age in good general health.
* Primary axillary hyperhidrosis of at least 6 months duration.
* Hyperhidrosis Disease Severity Score (HDSS) of 3 or 4 at baseline.
* Gravimetric test at baseline indicating at least 100mg of axillary sweat production in a 5 min period.
* Use of a medically appropriate contraceptive method.

Exclusion Criteria:

* Prior axillary use of botulinum toxin within 2 years of study entry.
* Prior iontophoresis treatment for axillary hyperhidrosis within 12 weeks of study entry.
* Prior surgical procedures for hyperhidrosis or surgical procedures in the axillary areas for any reason.
* Use of anticholinergic treatment, beta-blocker, alpha-adrenergic or other prescription treatment for hyperhidrosis.
* History of diabetes mellitus, thyroid disease, malignancy, glaucoma, intestinal obstructive or motility disease, obstructive uropathy, myasthenia gravis, prostate hypertrophy, neurological conditions or cardiac abnormalities.
* Known condition that may cause hyperhidrosis.
* Use of an investigational drug within 30 days prior to entry into this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Percent change in the gravimetrically measured sweat production from baseline | Week 2

SECONDARY OUTCOMES:
Absolute change in the gravimetrically measured sweat production from baseline | Week 2
Proportion of subjects who have a minimum of 2-grade improvement in HDSS from baseline. | Week 2
Proportion of subjects who have a minimum of 1-grade improvement in HDSS from baseline | Week 2